CLINICAL TRIAL: NCT02268994
Title: A Phase 3 Study of KRX-0502 (Ferric Citrate) for the Treatment of Iron Deficiency Anemia (IDA) in Adult Subjects With Non-Dialysis Dependent (NDD) Chronic Kidney Disease
Brief Title: KRX-0502 (Ferric Citrate) for the Treatment of IDA in Adult Subjects With NDD-CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KRX-0502-306
Record Dates: First submitted 2014-10-11; First posted 2014-10-20 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: ferric citrate; Chronic kidney disease; Anemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — ferric citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KRX-0502 (ferric citrate) (Experimental): 1 g of KRX-0502 (ferric citrate) containing approximately 210 mg of ferric iron
  Interventions: Drug: ferric citrate
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ferric citrate — 1 g ferric citrate containing approximately 210 mg of ferric iron
  Other Names: KRX-0502
  Arms: KRX-0502 (ferric citrate)
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
a 24-week phase 3, multi-center clinical trial, comprised of a 16-week, randomized, double-blind, placebo-controlled period ("Randomized Period"), followed by an 8-week open-label safety extension period, where all subjects receive KRX-0502 (ferric citrate) ("Extension Period").

DETAILED DESCRIPTION:
a 24-week phase 3, multi-center clinical trial, comprised of a 16-week, randomized, double-blind, placebo-controlled period ("Randomized Period"), followed by an 8-week open-label safety extension period, where all subjects receive KRX-0502 (ferric citrate) ("Extension Period"). The study will consist of 14 clinic visits over a period of 24 weeks. There will be a screening period of up to 14 days; Approximately 230 subjects will be randomized into the Randomized Period in a 1:1 ratio to receive either KRX-0502 or matching placebo, at baseline

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-lactating women with negative serum pregnancy test (for women of child-bearing potential) at Screening
2. Age ≥18 years
3. CKD with Estimated Glomerular Filtration Rate (eGFR) <60 mL/min at Screening using the 4-variable Modification of Diet in Renal Disease (MDRD) equation (with a limit of up to 20% of the target randomization of 230 subjects with eGFR <15 mL/min)
4. Patients who were intolerant of or have had an inadequate therapeutic response to oral iron supplements (in the opinion of the investigator)
5. Hgb ≥ 9.0 g/dL and ≤11.5 g/dL at Screening
6. Serum ferritin ≤200 ng/mL and Transferrin Saturation (TSAT) ≤25% at Screening
7. Serum Intact Parathyroid Hormone (iPTH) ≤600 pg/mL at Screening
8. Must consume a minimum of 2 meals per day
9. Willing and able to give written informed consent

Exclusion Criteria:

1. Serum phosphate <3.5 mg/dL at Screening
2. Liver enzymes (ALT/AST) >X3 times upper limit of normal at Screening
3. Symptomatic gastrointestinal bleeding or inflammatory bowel disease within 12 weeks prior to Screening
4. Evidence of acute kidney injury or requirement for dialysis within 12 weeks prior to Screening
5. Scheduled kidney transplant or initiation of dialysis planned within 24 weeks of Screening
6. IV iron administered within 4 weeks prior to Screening
7. Erythropoiesis-stimulating agent (ESA) administered within 4 weeks prior to Screening
8. Blood transfusion within 4 weeks prior to Screening
9. Receipt of any investigational drug within 4 weeks prior to Screening
10. Cause of anemia other than iron deficiency or chronic kidney disease
11. Malignancy (except non-melanoma skin cancer or disease-free for ≥2 years after curative therapy)
12. History of hemochromatosis
13. Active drug or alcohol dependence or abuse (excluding tobacco use or medicinal marijuana) within the 12 months prior to Screening or evidence of such abuse (in the opinion of the PI)
14. Subjects with known allergic reaction to previous oral iron therapy
15. Previous intolerance to oral ferric citrate
16. Psychiatric disorder that interferes with the subject's ability to comply with the study protocol
17. Planned surgery or hospitalization (anticipated to last >72 hours) during the randomized period of the trial other than dialysis access related surgery.
18. Any other medical condition that, in the opinion of the PI, renders the subject unable to or unlikely to complete the trial or that would interfere with optimal participation in the trial or produce significant risk to the subject
19. Inability to cooperate with study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Block, MD, Study Chair — Denver Nephrology; Glenn Chertow, MD, Study Chair — Division of Nephrology at Stanford University School of Medicine; Steven Fishbane, MD, Study Chair — Kidney Disease and Hypertension at North Shore University Hospital/Long Island Jewish Medical Center
Locations (36):
- United States (36):
  - AKDHC Medical Research Services, LLC, Phoenix, Arizona
  - Southwest Kidney Institute, Tempe, Arizona
  - California Renal Research, Glendale, California
  - Southern California Medical Research Center, La Palma, California
  - Academic Medical Research Institute, Inc, Los Angeles, California
  - Apex Research of Riverside, Riverside, California
  - Capital Nephrology Medical Group, Sacramento, California
  - La Jolla Clinical Research, Inc, San Diego, California
  - California Institute of Renal Research, San Diego, California
  - Denver Nephrology, Denver, Colorado
  - Creekside Medical Research, DeLand, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Pines Clinical Research, Inc, Pembroke Pines, Florida
  - Kidney Care Associates, LLC, Augusta, Georgia
  - Renal Physicians of Georgia, PC, Macon, Georgia
  - Pacific Renal Research Institute, Meridian, Idaho
  - Advanced Renal Care, Evergreen Park, Illinois
  - Kansas Nephrology Research Institute, Wichita, Kansas
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Western New England Renal & Transplant Associates, Springfield, Massachusetts
  - Renaissance Renal Research, Detroit, Michigan
  - Michigan Kidney Consultants, PC, Pontiac, Michigan
  - Clinical Research Consultants, Kansas City, Missouri
  - Lincoln Nephrology & Hypertension, Lincoln, Nebraska
  - Sierra Nevada Nephrology Asoociates, Reno, Nevada
  - Mountain Kidney & Hypertension Associates, Asheville, North Carolina
  - Metrolina Nephrology, Charlotte, North Carolina
  - Research Management, Inc, Austin, Texas
  - Research Management, Inc., Austin, Texas
  - TAD Clinical Research, Lufkin, Texas
  - Kidney & Hypertension Specialists, San Antonio, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - San Antonio Kidney Disease Center, San Antonio, Texas
  - Mendez Center for Clinical Research, Alexandria, Virginia
  - Nephrology Associates of Northern VA, Inc., Fairfax, Virginia
  - Peninsula Kidney Associates, Hampton, Virginia

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 randomized subject was excluded because they did not receive study drug and were excluded from the safety population.
Period: Overall Study
Arm/Group | KRX-0502 (Ferric Citrate) | Placebo
Started | 117 | 116
Completed | 86 | 81
Not Completed | 31 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KRX-0502 (Ferric Citrate) | Placebo | Total
Number analyzed (Participants) | 117 | 116 | 233
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 48 | 96
  >=65 years | 69 | 68 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (11.15) | 65.2 (13.08) | 65.4 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 71 | 147
  Male | 41 | 45 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 24 | 53
  Not Hispanic or Latino | 88 | 92 | 180
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 31 | 69
  White | 78 | 82 | 160
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving an Increase in Hemoglobin of ≥1.0 g/dL at Any Time Point Between Baseline and the End of the 16-week Randomized Period
Description: Efficacy analyses were performed for the Intention-to-treat (ITT) population, the population consisted of all subjects who were randomized, had a baseline laboratory value, took at least 1 dose of study drug, and had at least 1 post-baseline laboratory assessment during the randomized period.
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Groups:
- KRX-0502 (Ferric Citrate): 1 g KRX-0502 (ferric citrate) containing approximately 210 mg of ferric iron
  ferric citrate: 1 gr ferric citrate containing approximately 210 mg of ferric iron
Arm/Group | KRX-0502 (Ferric Citrate) | Placebo
Number analyzed (Participants) | 117 | 115
Participants | 61 | 22

2. Secondary Outcome: Mean Change in Hemoglobin (Hgb) at the End of 16 Weeks Minus Baseline
Description: The difference of Hgb at 16 weeks compared to the Hgb value at the time of study entry.
Time Frame: Baseline and week 16
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | KRX-0502 (Ferric Citrate) | Placebo
Number analyzed (Participants) | 117 | 115
g/dL | 0.39 (0.054) | -0.14 (0.056)

3. Secondary Outcome: Mean Change in Transferrin Saturation (TSAT) at the End of 16 Weeks Minus Baseline
Description: The difference of TSAT at 16 weeks compared to the TSAT value at the time of study entry was averaged.
Time Frame: Baseline and week 16
Measure: Least Squares Mean (Standard Error); unit: % saturation
Groups:
- KRX-0502 (Ferric Citrate): 1 g KRX-0502 (ferric citrate) containing approximately 210 mg of ferric iron
  ferric citrate: 1 g ferric citrate containing approximately 210 mg of ferric iron
Arm/Group | KRX-0502 (Ferric Citrate) | Placebo
Number analyzed (Participants) | 117 | 115
% saturation | 10.9 (0.65) | -1.3 (0.67)

4. Secondary Outcome: Mean Change in Ferritin at the End of 16 Weeks Minus Baseline
Description: The difference of ferritin at 16 weeks compared to the ferritin value at the time of study entry.
Time Frame: Baseline and week 16
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Groups:
- KRX-0502 (Ferric Citrate): 1 gr of KRX-0502 (ferric citrate) containing approximately 210 mg of ferric iron
  ferric citrate: 1 g ferric citrate containing approximately 210 mg of ferric iron
Arm/Group | KRX-0502 (Ferric Citrate) | Placebo
Number analyzed (Participants) | 117 | 115
ng/mL | 68.1 (3.99) | -6.1 (4.10)

5. Secondary Outcome: Percentage of Subjects Experiencing a Sustained Treatment Effect on Hemoglobin (Hgb)
Description: Proportion of subjects that continued to maintain an increase in Hgb over a 4 week period, provided they had an increase of at least 1.0 g/dL during that 4-week period
Time Frame: Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | KRX-0502 (Ferric Citrate) | Placebo
Number analyzed (Participants) | 117 | 115
Participants | 57 | 17

6. Secondary Outcome: Mean Change in Serum Phosphate at the End of 16 Weeks Minus Baseline
Description: The difference of serum phosphate at 16 weeks compared to the serum phosphate value at the time of study entry.
Time Frame: Baseline and week 16
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | KRX-0502 (Ferric Citrate) | Placebo
Number analyzed (Participants) | 117 | 115
mg/dL | -0.28 (0.036) | -0.14 (0.037)

ADVERSE EVENTS:
Time Frame: 16 Week Randomized Period
Arm/Group | KRX-0502 (Ferric Citrate) | Placebo
All-Cause Mortality (participants affected / at risk) | 2/117 | 0/116
Serious Adverse Events (participants affected / at risk) | 14/117 | 13/116
Other Adverse Events (participants affected / at risk) | 61/117 | 41/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KRX-0502 (Ferric Citrate) (N=117) | Placebo (N=116)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 2
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Necrosis (General disorders) | 0 | 1
Cholangitis Acute (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Clostridium Difficle Colitis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Abscess Limb (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Urinary Tract Infection Fungal (Infections and infestations) | 1 | 0
Celluitis (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural Nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural Vomiting (Injury, poisoning and procedural complications) | 1 | 0
Blood Glucose Increased (Investigations) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Metabolic Encephalopathy (Nervous system disorders) | 2 | 0
Status Epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 3 | 2
Renal Failure Chronic (Renal and urinary disorders) | 1 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Toe Amputation (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KRX-0502 (Ferric Citrate) (N=117) | Placebo (N=116)
Diarrhoea (Gastrointestinal disorders) | 24 | 19
Constipation (Gastrointestinal disorders) | 22 | 15
Faeces Discoloured (Gastrointestinal disorders) | 17 | 0
Nausea (Gastrointestinal disorders) | 13 | 3
Abdominal Pain (Gastrointestinal disorders) | 7 | 2
Fatigue (General disorders) | 0 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 4
Hypertension (Vascular disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days